CLINICAL TRIAL: NCT01687777
Title: Treatment of Rotator Cuff Tears Using Autologous Bone Marrow Mensenchymal Stem Cell Transplantation.
Brief Title: Mensenchymal Stem Cell (MSC) Included in OrthADAPT Membrane for Rotator Cuff Tears Repair
Acronym: msctendonrep
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Benjamin Fernandez Gutierrez, Rheumatologist, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC07/90208; 2007-007630-19 (EudraCT Number)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Disease
Keywords: Supraspinatus tendon; Mesenchymal stem cells; OrthADAPT; Rotator cuff
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesenchymal stem cells (MSCs) (Active Comparator): Mesenchymal stem cells with a collagen type I membrane (OrthoADAPT)
  Interventions: Biological: Mesenchymal Stem Cells (MSCs)
- OrthADAPT (Placebo Comparator): Membrane of collagen type I (OrthoADAPT)
  Interventions: Biological: OrthADAPT

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSCs) — 20.000.000 autologous MSCs included in the OrthADAPT membrane. Single dosage.
  Arms: Mesenchymal stem cells (MSCs)
Biological: OrthADAPT
  Arms: OrthADAPT

SUMMARY:
Surgical reconstructive procedures for rotator cuff tears present a number of limitations. The few studies in which the repair integrity is evaluated, have shown the existence of a high rate of reruptures in spite of the fact that the functional results obtained short-term are satisfactory. Morphologic analysis from the sutures, after different follow-up periods, has not shown satisfactory results.

Thus, the purpose of the current study was to test the hypotheses that mesenchymal stem cells (MSCs) included in a membrane into rotator cuff tears improves, the radiograms and the function compared to cell-free tendon defect treatment.

DETAILED DESCRIPTION:
The investigators will include: Patients with massive tears from the supraspinatus tendon, in which reconstructive surgery is indicated. Patients will be randomly stratified into two groups.

The first group will receive autologous MSCs transplantation included in a collagen type I membrane (OrthADAPT) and the second group will serve as cell-free controls.

The surgical procedure will be performed by arthroscopic and/or combined technique: arthroscopic subacromial decompression and mini-open rotator cuff repair. The OrthADAPT-cells composite will be put on the sutured area. The radiograms and function will be assessed by independently observers, who will no have knowledge of the study group from which they will have been obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subject providing informed consent.
* Comprised subject male/female aged 55-80.
* Subject has a supraspinatus tendon rupture.
* Subject has an unilateral injury.
* Rupture is enough to need medical assistance.
* Subject has an conventional medical treatment fail at least 3 months.
* Subject has a "reparable" injury according to Goutallier´s criteria.

Exclusion Criteria:

* Subject has a prior clinical history of arthritis, diabetes or inflammatory disease.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Constant Shoulder Score | up to 1 year

SECONDARY OUTCOMES:
Nuclear Magnetic Resonance (RMN) | 6 months, one year

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Fernandez-Gutierrez, MD, PhD, Principal Investigator — Hospital Universitario Clinico San Carlos; Pilar Tornero-Esteban, Bs, PhD, Study Director — Hospital Universitario Clinico San Carlos
Locations (1):
- Hospital Universitario Clinico San Carlos, Madrid, Madrid, Spain

REFERENCES:
- [Background] Awad HA, Butler DL, Boivin GP, Smith FN, Malaviya P, Huibregtse B, Caplan AI. Autologous mesenchymal stem cell-mediated repair of tendon. Tissue Eng. 1999 Jun;5(3):267-77. doi: 10.1089/ten.1999.5.267. PMID 10434073
- [Background] Awad HA, Boivin GP, Dressler MR, Smith FN, Young RG, Butler DL. Repair of patellar tendon injuries using a cell-collagen composite. J Orthop Res. 2003 May;21(3):420-31. doi: 10.1016/S0736-0266(02)00163-8. PMID 12706014
- [Background] Barber FA, Aziz-Jacobo J. Biomechanical testing of commercially available soft-tissue augmentation materials. Arthroscopy. 2009 Nov;25(11):1233-9. doi: 10.1016/j.arthro.2009.05.012. Epub 2009 Oct 2. PMID 19896044
- [Background] Bruder SP, Jaiswal N, Haynesworth SE. Growth kinetics, self-renewal, and the osteogenic potential of purified human mesenchymal stem cells during extensive subcultivation and following cryopreservation. J Cell Biochem. 1997 Feb;64(2):278-94. doi: 10.1002/(sici)1097-4644(199702)64:23.0.co;2-f. PMID 9027588
- [Background] Bruder SP, Kraus KH, Goldberg VM, Kadiyala S. The effect of implants loaded with autologous mesenchymal stem cells on the healing of canine segmental bone defects. J Bone Joint Surg Am. 1998 Jul;80(7):985-96. doi: 10.2106/00004623-199807000-00007. PMID 9698003
- [Background] Caplan AI. Mesenchymal stem cells. J Orthop Res. 1991 Sep;9(5):641-50. doi: 10.1002/jor.1100090504. PMID 1870029
- [Background] Caplan AI. The mesengenic process. Clin Plast Surg. 1994 Jul;21(3):429-35. PMID 7924141
- [Background] Caplan AI. Review: mesenchymal stem cells: cell-based reconstructive therapy in orthopedics. Tissue Eng. 2005 Jul-Aug;11(7-8):1198-211. doi: 10.1089/ten.2005.11.1198. PMID 16144456
- [Background] Cofield RH, Parvizi J, Hoffmeyer PJ, Lanzer WL, Ilstrup DM, Rowland CM. Surgical repair of chronic rotator cuff tears. A prospective long-term study. J Bone Joint Surg Am. 2001 Jan;83(1):71-7. doi: 10.2106/00004623-200101000-00010. PMID 11205861
- [Background] Djurasovic M, Marra G, Arroyo JS, Pollock RG, Flatow EL, Bigliani LU. Revision rotator cuff repair: factors influencing results. J Bone Joint Surg Am. 2001 Dec;83(12):1849-55. doi: 10.2106/00004623-200112000-00013. PMID 11741065
- [Background] Galatz LM, Ball CM, Teefey SA, Middleton WD, Yamaguchi K. The outcome and repair integrity of completely arthroscopically repaired large and massive rotator cuff tears. J Bone Joint Surg Am. 2004 Feb;86(2):219-24. doi: 10.2106/00004623-200402000-00002. PMID 14960664
- [Background] Gimbel JA, Van Kleunen JP, Lake SP, Williams GR, Soslowsky LJ. The role of repair tension on tendon to bone healing in an animal model of chronic rotator cuff tears. J Biomech. 2007;40(3):561-8. doi: 10.1016/j.jbiomech.2006.02.010. Epub 2006 Apr 4. PMID 16600252
- [Background] Goutallier D, Postel JM, Gleyze P, Leguilloux P, Van Driessche S. Influence of cuff muscle fatty degeneration on anatomic and functional outcomes after simple suture of full-thickness tears. J Shoulder Elbow Surg. 2003 Nov-Dec;12(6):550-4. doi: 10.1016/s1058-2746(03)00211-8. PMID 14671517
- [Background] Harryman DT 2nd, Mack LA, Wang KY, Jackins SE, Richardson ML, Matsen FA 3rd. Repairs of the rotator cuff. Correlation of functional results with integrity of the cuff. J Bone Joint Surg Am. 1991 Aug;73(7):982-9. PMID 1874784
- [Background] Jaiswal N, Haynesworth SE, Caplan AI, Bruder SP. Osteogenic differentiation of purified, culture-expanded human mesenchymal stem cells in vitro. J Cell Biochem. 1997 Feb;64(2):295-312. PMID 9027589
- [Background] Johnson W, Inamasu J, Yantzer B, Papangelou C, Guiot B. Comparative in vitro biomechanical evaluation of two soft tissue defect products. J Biomed Mater Res B Appl Biomater. 2007 Apr 5. doi: 10.1002/jbm.b.30816. Online ahead of print. PMID 17415772
- [Background] Jost B, Pfirrmann CW, Gerber C, Switzerland Z. Clinical outcome after structural failure of rotator cuff repairs. J Bone Joint Surg Am. 2000 Mar;82(3):304-14. doi: 10.2106/00004623-200003000-00002. PMID 10724223
- [Background] Mansilla E, Marin GH, Sturla F, Drago HE, Gil MA, Salas E, Gardiner MC, Piccinelli G, Bossi S, Salas E, Petrelli L, Iorio G, Ramos CA, Soratti C. Human mesenchymal stem cells are tolerized by mice and improve skin and spinal cord injuries. Transplant Proc. 2005 Jan-Feb;37(1):292-4. doi: 10.1016/j.transproceed.2005.01.070. PMID 15808623
- [Background] Pillow RP, Epstein RB, Buckner CD, Giblett ER, Thomas ED. Treatment of bone-marrow failure by isogeneic marrow infusion. N Engl J Med. 1966 Jul 14;275(2):94-7. doi: 10.1056/NEJM196607142750209. No abstract available. PMID 5327813
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Prickett WD, Teefey SA, Galatz LM, Calfee RP, Middleton WD, Yamaguchi K. Accuracy of ultrasound imaging of the rotator cuff in shoulders that are painful postoperatively. J Bone Joint Surg Am. 2003 Jun;85(6):1084-9. doi: 10.2106/00004623-200306000-00016. PMID 12784007
- [Background] Saito T, Dennis JE, Lennon DP, Young RG, Caplan AI. Myogenic Expression of Mesenchymal Stem Cells within Myotubes of mdx Mice in Vitro and in Vivo. Tissue Eng. 1995 Winter;1(4):327-43. doi: 10.1089/ten.1995.1.327. PMID 19877897
- [Background] Romeo AA, Hang DW, Bach BR Jr, Shott S. Repair of full thickness rotator cuff tears. Gender, age, and other factors affecting outcome. Clin Orthop Relat Res. 1999 Oct;(367):243-55. PMID 10546622
- [Background] Smith RK, Korda M, Blunn GW, Goodship AE. Isolation and implantation of autologous equine mesenchymal stem cells from bone marrow into the superficial digital flexor tendon as a potential novel treatment. Equine Vet J. 2003 Jan;35(1):99-102. doi: 10.2746/042516403775467388. No abstract available. PMID 12553472
- [Background] Wakitani S, Goto T, Pineda SJ, Young RG, Mansour JM, Caplan AI, Goldberg VM. Mesenchymal cell-based repair of large, full-thickness defects of articular cartilage. J Bone Joint Surg Am. 1994 Apr;76(4):579-92. doi: 10.2106/00004623-199404000-00013. PMID 8150826
- [Background] Yamaguchi K, Levine WN, Marra G, Galatz LM, Klepps S, Flatow EL. Transitioning to arthroscopic rotator cuff repair: the pros and cons. Instr Course Lect. 2003;52:81-92. PMID 12690842